CLINICAL TRIAL: NCT02999243
Title: Development of an HIV Self-testing Intervention to Reduce HIV Risks Among MSM: Taking the Guess Out of Seroguessing
Brief Title: Development of an HIV Self-testing Intervention
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: IRB expired, PI no longer at institution.
Sponsor: University of California, San Francisco (Other)
Collaborators: Jiangsu Provincial Center for Diseases Control and Prevention, China (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1R34MH109359 (NIH)
Record Dates: First submitted 2016-12-14; First posted 2016-12-21 (Estimated); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: HIV Serosorting
MeSH Terms: conditions — HIV Serosorting

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIV self-testing (Experimental): HIV self-testing kits plus harm reduction education materials will be offered to the intervention group.
  Interventions: Behavioral: HIV self-testing; Behavioral: Harm reduction education
- Education (Placebo Comparator): Harm reduction educational materials will be offered to the control group.
  Interventions: Behavioral: Harm reduction education

INTERVENTIONS:
Behavioral: HIV self-testing — The intervention group will be offered HIV self-testing kits for testing HIV status
  Arms: HIV self-testing
Behavioral: Harm reduction education — Both arms will receive harm reduction education

SUMMARY:
This randomized controlled trial (RCT) evaluates whether HIV self-testing (HIVST) facilitates sexual harm reduction and reduces HIV transmission among HIV-negative MSM in China.The intervention group will be offered HIVST kits plus harm reduction education, and followed 9 month, while the control group will receive harm reduction educational material only.

DETAILED DESCRIPTION:
The HIV epidemic in China is now concentrated among men who have sex with men (MSM), who account for a third of new HIV infections. Despite strengthened prevention efforts and increased availability of HIV testing in the country, testing rates are low and condomless sex is common among Chinese MSM. Globally, condomless sex among MSM, particularly with primary partners, is also ubiquitous. To reduce HIV transmission risks in the context of condomless sex, MSM communities have adopted a range of sexual harm reduction strategies (i.e., seroadaptive behaviors). Essential to the effectiveness of these strategies is accurate knowledge of HIV status within the partnership. This necessitates frequent HIV testing and mutual HIV status disclosure. However, significant proportions of MSM have never tested or not recently tested and are unaware of their own and their partner's HIV status, especially in settings where sexual minorities are stigmatized. Among Chinese MSM, their ability to successfully use these harm reduction strategies is severely limited by low levels of HIV testing and disclosure efficacy. As a result, many Chinese MSM make unreliable assumptions about their own and their partners' serostatus (i.e., seroguessing), resulting in risky condomless sex. As many of these men do not access facility-based testing, new and emerging HIV testing options must be expanded to help these men make informed decisions about sexual risk and harm reduction. HIV self-testing (HIVST) offers a promising prevention strategy to reach more untested Chinese MSM, increase testing frequency, and serve as a valuable prevention tool to assist harm reduction. The investigators propose to determine the feasibility and preliminary efficacy of an HIVST intervention in facilitating sexual harm reduction and reducing HIV transmission among MSM in Nanjing, China. The investigators will: 1) conduct participant observation (N = 20) and cognitive interviews (N=10) to determine what information and support is needed for MSM to use HIVST safely and practice sexual harm reduction responsibly; and 2) recruit and enroll 400 high-risk HIV-negative MSM into a RCT where the intervention group will be offered HIVST kits plus harm reduction education and followed over a 9-month period to determine whether the intervention increases uptake and frequency of testing in partnership, improves disclosure and awareness of partners' HIV status, and therefore facilitates sexual harm reduction and reduces HIV transmission. Expanding HIV testing among key populations is a priority for HIV prevention worldwide. Innovative strategies are needed to encourage MSM to seek HIV testing while taking into consideration existing paradigms of community-originated and driven harm reduction strategies. As HIVST is being introduced to different settings and becoming more accessible, findings from this proposed study will provide vital information on current patterns of seroadaptation and HIVST use; identify what is needed to promote HIVST's proper use for harm reduction and linkage to HIV/STI care, and whether HIVST can improve the accuracy of harm reduction strategies.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years or older;
* born male;
* currently residing in Nanjing and planning to stay as a resident during the study period;
* speaks either Mandarin or the local dialect;
* confirmed HIV negative through HIV rapid testing;
* have had condomless anal sex with a man in the past six months

Exclusion Criteria:

-

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2018-05-21 (Actual); Study Completion 2018-05-21 (Actual)

PRIMARY OUTCOMES:
Change in participants' HIV testing uptake | Baseline and 9-month
  Change in proportion of participants being tested for HIV

SECONDARY OUTCOMES:
Change in partners' HIV testing uptake | Baseline and 9-month
  Change in proportion of participants' partners who tested for HIV
Questionnaire to assess change in awareness of partner's HIV status | Baseline and 9-month
  Change in proportion of participants' who report that they are aware of their partners' HIV status
Questionnaire to assess change in self-reported sexually transmitted infection (STI) symptoms | Baseline and 9-month
  Change in proportion of participants who report symptoms of STIs
Incident HIV infection | Baseline and 9-month

CONTACTS AND LOCATIONS:
Overall Officials: Chongyi Wei, DrPH, Principal Investigator — University of California, San Francisco
Locations (1):
- Jiangsu Provincial Center for Disease Control and Prevention, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li D, Li S, Liu Y, Gao Y, Yu M, Yang X, Li Q, Jiang S, Zhou Z, Zhang Z, Yan L, Jiang G, Xiao D, Pan SW, Luo F, Ruan Y, Shao Y. HIV incidence among men who have sex with men in Beijing: a prospective cohort study. BMJ Open. 2012 Nov 19;2(6):e001829. doi: 10.1136/bmjopen-2012-001829. Print 2012. PMID 23166133
- [Background] Wang QQ, Chen XS, Yin YP, Liang GJ, Zhang RL, Jiang N, Huan XP, Yang B, Liu Q, Zhou YJ, Wang BX. HIV prevalence, incidence and risk behaviours among men who have sex with men in Yangzhou and Guangzhou, China: a cohort study. J Int AIDS Soc. 2014 Aug 6;17(1):18849. doi: 10.7448/IAS.17.1.18849. eCollection 2014. PMID 25103308
- [Background] Xu JJ, Zhang M, Brown K, Reilly K, Wang H, Hu Q, Ding H, Chu Z, Bice T, Shang H. Syphilis and HIV seroconversion among a 12-month prospective cohort of men who have sex with men in Shenyang, China. Sex Transm Dis. 2010 Jul;37(7):432-9. doi: 10.1097/OLQ.0b013e3181d13eed. PMID 20375928
- [Background] Yan H, Yang H, Zhao J, Wei C, Li J, Huan X, Zhang M, Raymond HF, McFarland W. Long-chain peer referral of men who have sex with men: a novel approach to establish and maintain a cohort to measure HIV incidence, Nanjing, China. J Acquir Immune Defic Syndr. 2012 Feb 1;59(2):177-84. doi: 10.1097/QAI.0b013e318239c947. PMID 21992923
- [Background] Chow EP, Iu KI, Fu X, Wilson DP, Zhang L. HIV and sexually transmissible infections among money boys in China: a data synthesis and meta-analysis. PLoS One. 2012;7(11):e48025. doi: 10.1371/journal.pone.0048025. Epub 2012 Nov 29. PMID 23209551
- [Background] Snowden JM, Wei C, McFarland W, Raymond HF. Prevalence, correlates and trends in seroadaptive behaviours among men who have sex with men from serial cross-sectional surveillance in San Francisco, 2004-2011. Sex Transm Infect. 2014 Sep;90(6):498-504. doi: 10.1136/sextrans-2013-051368. Epub 2014 Mar 31. PMID 24687128
- [Background] Eaton LA, Kalichman SC, O'Connell DA, Karchner WD. A strategy for selecting sexual partners believed to pose little/no risks for HIV: serosorting and its implications for HIV transmission. AIDS Care. 2009 Oct;21(10):1279-88. doi: 10.1080/09540120902803208. PMID 20024704
- [Background] Xia Q, Molitor F, Osmond DH, Tholandi M, Pollack LM, Ruiz JD, Catania JA. Knowledge of sexual partner's HIV serostatus and serosorting practices in a California population-based sample of men who have sex with men. AIDS. 2006 Oct 24;20(16):2081-9. doi: 10.1097/01.aids.0000247566.57762.b2. PMID 17053354
- [Background] Mitchell JW, Horvath KJ. Factors associated with regular HIV testing among a sample of US MSM with HIV-negative main partners. J Acquir Immune Defic Syndr. 2013 Dec 1;64(4):417-23. doi: 10.1097/QAI.0b013e3182a6c8d9. PMID 23933766
- [Background] Centers for Disease Control and Prevention (CDC). Prevalence and awareness of HIV infection among men who have sex with men --- 21 cities, United States, 2008. MMWR Morb Mortal Wkly Rep. 2010 Sep 24;59(37):1201-7. PMID 20864920
- [Background] He N, Detels R. The HIV epidemic in China: history, response, and challenge. Cell Res. 2005 Nov-Dec;15(11-12):825-32. doi: 10.1038/sj.cr.7290354. PMID 16354555
- [Background] Gari S, Doig-Acuna C, Smail T, Malungo JR, Martin-Hilber A, Merten S. Access to HIV/AIDS care: a systematic review of socio-cultural determinants in low and high income countries. BMC Health Serv Res. 2013 May 28;13:198. doi: 10.1186/1472-6963-13-198. PMID 23714167
- [Derived] Wei C, Yan L, Li J, Su X, Lippman S, Yan H. Which user errors matter during HIV self-testing? A qualitative participant observation study of men who have sex with men (MSM) in China. BMC Public Health. 2018 Sep 10;18(1):1108. doi: 10.1186/s12889-018-6007-3. PMID 30200905